CLINICAL TRIAL: NCT02289053
Title: Prevalence and Topography of Adenomas in 40-49 Year Old Patients With a Family History of Colon Cancer
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Philip Schoenfeld, Professor of Medicine, University of Michigan
Other Study IDs: K24-DK; 1K24DK084208 (NIH)
Record Dates: First submitted 2014-02-26; First posted 2014-11-13 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer; Colon Polyps; Adenomatous Polyp of Colon
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Positive Family History: Eligible participants with a family history of colorectal cancer or polyps will be grouped into the "subjects" group.
- Average Risk Patients: Eligible participants without a family history of colorectal cancer or polyps will be grouped into the "control" group.

SUMMARY:
Conflicting guideline recommendations for screening colonoscopy result due to scant data upon which to develop appropriate recommendations. No previous study has compared the prevalence of advanced adenomas or adenomas (any size) among 40-49 year old individuals with a first degree relative (FDR) with colorectal cancer (CRC) versus 40-49 year old average risk individuals with no family history of CRC. The purpose of this study is to determine the prevalence of colon adenomas in 40-49 year old individuals and identify risk factors associated with the presence of advanced adenomas. This data will provide evidence to determine appropriate colon cancer screening guidelines in 40-49 year old persons with a family history of colon polyps or colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 40-49 year old asymptomatic men and women referred for colorectal cancer screening with a family history of CRC in a first degree relative;
* 40-49 year old asymptomatic men and women referred for colorectal cancer screening with a family history of polyps in a first degree relative;
* 40-49 year old men and women without a family history of CRC or polyps in a first degree relative who are referred for colonoscopy to evaluate scant hematochezia characterized as red blood on toilet tissue after wiping or small droplets of blood on stool or in toilet water after evacuating stool, abdominal discomfort or altered bowel habits characterized as constipation or diarrhea.

Exclusion Criteria:

* Personal history of iron deficiency anemia within six months of referral;
* Personal history of iron deficiency without anemia within six months of referral;
* Personal history of (+) FOBT within one year of referral;
* Personal history of previous colonoscopy or barium enema within the past 10 years;
* Personal history of previous flexible sigmoidoscopy in the past 5 years;
* Personal history of adenoma, colorectal cancer, inflammatory bowel disease, HNPCC, or familial adenomatous polyposis (FAP);
* Unintentional weight loss > 10 lbs within the previous six months;
* Individuals with family history of CRC AND scant hematochezia;
* Inability to speak and read English.

Ages: 40 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants are recruited from the endoscopy units of the participating study sites prior to their colonoscopy procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1623 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of advanced adenomas among 40-49 year old individuals with and without a family history of colorectal cancer | Data analysis will begin September 2014 for a duration of three months.
  The outcome will be assessed after the completion of patient recruitment at all locations in August 2014. Advanced adenomas are defined as greater than or equal to 10 mm (1 cm). The presence of adenomas is determined be reviewing patient medical records and pathology reports.

SECONDARY OUTCOMES:
Absolute prevalence of advanced adenomas in 40-49 year olds with a family history of colorectal cancer | Data analysis will begin September 2014 for a duration of three months.
  The outcome will be assessed after the completion of patient recruitment at all locations in August 2014. Advanced adenomas are defined as greater than or equal to 10 mm (1 cm). The presence of adenomas is determined be reviewing patient medical records and pathology reports.
Absolute prevalence of advanced adenomas in 40-49 year old individuals with a family history of colorectal polyps | Data analysis will begin September 2014 for a duration of three months.
  The outcome will be assessed after the completion of patient recruitment at all locations in August 2014. Advanced adenomas are defined as greater than or equal to 10 mm (1 cm). The presence of adenomas is determined be reviewing patient medical records and pathology reports.

OTHER OUTCOMES:
Risk factors associated with the presence of advanced adenomas | Data analysis will begin September 2014 for a duration of three months.
  Logistic regression will be used to determine if specific risk factors are associated with the risk of adenomas in 40-49 year old individuals. Data will be collected from patient surveys and medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Schoenfeld, MD, Principal Investigator — University of Michigan
Locations (6):
- United States (6):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Ann Arbor VA Healthcare System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center, Detroit, Michigan
  - Huron Gastro, Ypsilanti, Michigan
  - Durham VA Medical Center, Durham, North Carolina